CLINICAL TRIAL: NCT07029555
Title: A Phase Ib, Open-label, Ascending Dose Study to Assess Safety, Tolerability and Pharmacokinetics of PIT565 in Participants With Rheumatoid Arthritis (RA)
Brief Title: An Ascending Dose Study of PIT565 in Participants With Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPIT565C12101
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
Keywords: PIT565; ascending dose; rheumatoid arthritis; B cells
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- PIT565 dose 1 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 2 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 3 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 4 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 5 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 6 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 7 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565
- PIT565 dose 8 (Experimental): Study treatment will be provided in vials as open-label participant specific supply.
  Interventions: Biological: PIT565

INTERVENTIONS:
Biological: PIT565 — Study treatment will be provided in vials as open-label participant specific supply.

SUMMARY:
The purpose of the study is to determine the safety, tolerability, and pharmacokinetics of PIT565, in participants with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
This is an open-label, uncontrolled study in participants with RA. PIT565 will be administered subcutaneously. The objective of the study is to assess the safety and efficacy of PIT565 in participants with RA.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study. Male and female patients, aged 18 to 75 years at screening, diagnosed with RA according to the 2010 ACR/EULAR or 1987 ACR classification at least 12 weeks prior to screening.
* Immunization (primary or from vaccinations) against pneumococcus, influenza, and COVID-19 infection at least 2 weeks prior to the first dosing. Local guidelines should be followed to determine requirement for vaccination (or booster), as well as the type and schedule of vaccination.

Exclusion Criteria:

• Any of the following cardiac conditions

1. Unstable angina, myocardial infarction, coronary artery bypass graft (CABG), or stroke within 6 months prior to screening
2. Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥ 2) or uncontrolled hypertension
3. Concomitant clinically significant cardiac arrhythmias, e.g., sustained ventricular tachycardia, and clinically significant second or third degree atrioventricular block without a pacemaker
4. History of familial long QT syndrome or known family history of Torsades-de- Pointes
5. Resting QTcF ≥ 450 msec (male) or ≥ 460 msec (female) at screening
6. Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-16 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 6 months
  Incidence and severity of AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of PIT565: Maximum serum Concentration [Cmax] | up to 6 months
  Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass x volume-1)
Pharmacokinetic parameters of PIT565: Area under serum concentration (AUC) | up to 6 months
  AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1).
Concentrations of anti-PIT565 antibodies | Baseline, up to 6 months
  To assess the immunogenicity (IG) of PIT565

CONTACTS AND LOCATIONS:
Locations (10):
- Novartis Investigative Site, CABA, Argentina
- Novartis Investigative Site, Sofia, Bulgaria
- Novartis Investigative Site, Beijing, China
- Germany (2):
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Leiden, South Holland, Netherlands
- Romania (2):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Bucharest
- Spain (2):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No